CLINICAL TRIAL: NCT03258047
Title: Novel Autologou CAR-T Therapy for Relapsed/Refractory B Cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Principal Investigator, Wenbin Qian, Doctor, First Affiliated Hospital of Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: lymphoma center Q002
Record Dates: First submitted 2017-08-20; First posted 2017-08-22 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T treatment (Experimental): In this group, patients will be treated with autologous CAR-T, and the safety and efficacy will be evaluated
  Interventions: Combination Product: CAR-T

INTERVENTIONS:
Combination Product: CAR-T — CAR-T is a novel technique for cancer treatent, it includes procedures of modifying patients' T cells outside the body and re-transfuse these cells back into the human body to fight against the cancer cells.

SUMMARY:
It's a single arm, open label prospective study, in which the safety and efficacy of autologous CAR-T are evaluated in refractory/relapsed B cell lymphoma patients.

Abbreviation: CAR-T: Chimeric Antigen Receptor T-Cell Immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years, male or female;
2. Karnofsky≥60%；
3. B cell lymphoma patients who are not available for the following treatment: autologous stem cell transplantation, allogeneic stem cell transplantation, or patients with short expected survival (less than 2 years).
4. Patients with CR2 or CR3 and no stem cell transplantation available due to age, disease condition, lack of donors or any other reasons.
5. Patients have had more than 2 combined chemotherapy regimens;
6. Creatinin <2.5mg/dL；ALT/AST level <3 times of the maximum of normal range; bilirubin<3mg/dL；
7. Proper venous condition for leukapheresis, no contraindication for leukapheresis;
8. Patient that could understand and is willing to sign the written consent;
9. Fertile female patient should be willing to take contraceptive measures.
10. Patient that is willing to follow up till at least 2 months after T cell re-transfusion.

Exclusion Criteria:

1. Patients who need ≥15mg prednisone daily due to any cause;
2. Patients with autoimmune disease and need immunosuppressor treatment;
3. Serum creatinin>2.5 mg/dL；serum AST >5 times of normal maximum; bilirubin >3 mg/Dl;
4. FEV1<2 L，diffusion capacity for carbon monoxide of lung (DLCO) <40%；
5. Cardiovascular abnormalities that fulfill any of the following: NYHA level III or IV congestive heart failure, severe clinical hypotention; uncontrollable carotid heart disease; or ejection fraction<35%；
6. Patients with HIV infection, active Hepatitis B or Hepatitis C infection;
7. Patients that have previously received gene therapy of any kind;
8. Obvious clinical encephalopathy or novel neuron function damage;
9. Patients with active infection;
10. Patients had biological treatment, immunotherapy or radiation therapy within 1 month prior to enrollment or are currently under these treatment;
11. Patients who had allergic history to agents of the similar structure as CAR-T;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-09-15 (Actual); Primary Completion 2019-01-13 (Actual); Study Completion 2019-07-30 (Estimated)

PRIMARY OUTCOMES:
complete remission rate | every 3 months until 20 months after the last patient's enrollment
  complete remission rate after treated by CAR-T therapy

SECONDARY OUTCOMES:
progression free survival | from the day of treatment to the date of first documented progression，up to 20 months after the last patient's enrollment
  from date of inclusion to date of progression, relapse, or death from any cause
overall survival | 20 months after the last patient's enrollment
  from the date of inclusion to date of death, irrespective of cause
adverse events | from the date of the start of treatment to 20 months after last patient's enrollment
  any unfavorable and unintended sign , symptom, or disease temporally associated with the use of a medical treatment or procedure that may or may not be considered related to the medical treatment or procedure
duration of the modified T cells by CAR-T in the patients | from the date of re-transfusison to 20 months after last patient's enrollment
  time from re-transfusion to date when the modified T cells become non-detectable.

CONTACTS AND LOCATIONS:
Locations (1):
- The first affiliated hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
All the data would be available on the corresponding website of the leading research center.